CLINICAL TRIAL: NCT06265506
Title: Assessing the Clinical and Cost-Effectiveness of a Virtual PEth-based Contingency Management for Adults With AUD
Brief Title: Virtual Incentive Treatment for Alcohol
Acronym: VITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Weill Medical College of Cornell University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael McDonell, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20320; R01AA031013 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-02-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking; Alcohol Abuse; Alcohol Dependence
Keywords: Contingency Management; Alcohol Abstinence; Adult; Biological Markers; Blood; Clinical effectiveness; Cognitive Therapy; Blood collection; Ethyl glucuronide; Health Care Costs; Heavy Drinking; Addictions Neuroclinical Assessment; Cognition; Incentives; Phosphatidylethanol; Incentive salience; Anhedonia; Longitudinal Studies; Prediction of Response to Therapy; Randomized Clinical Trial; Telehealth; Virtual Health; Video conference
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcohol Abstinence; Anhedonia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: We will test the efficacy of our CM model against an evidence-based online intervention, CBT4CBT, by randomizing participants to six months of:
  1. CBT4CBT and reinforcement for submitting blood samples (no requirement for abstinence) (Control Condition), or
  2. CBT4CBT and reinforcement for PEth tests that are consistent with alcohol abstinence (CM Condition).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Non-contingent Incentives + CBT4CBT) (Active Comparator): Participants will receive 8 weeks of Computer Based Training for Cognitive Behavioral Health (CBT4CBT). CBT4BCT is a self paced web-based program that uses videos and lessons to help people learn skills they can use to cut down or stop drinking. Participants will receive a $10 e-gift card for every PEth sample submitted within 48 hours of the visit regardless of the result. Participants will receive gift card incentives when they attend visits and provide blood samples (PEth Samples). Participants will submit PEth samples weekly for the first four weeks of the study, then every two weeks (weeks six, eight), then every four weeks (weeks 12,16, 20, 24), and at week 26. Each time they submit a PEth sample, they will receive gift cards equal to the average CM earnings during the previous month, resulting in total average earnings equivalent to the CM group. This group will receive incentives regardless of the results of their PEth tests.
  Interventions: Behavioral: Computer Based Training for Cognitive Behavioral Therapy for AUD (CBT4CBT)
- CM Condition (Contingency Management + CBT4CBT) (Experimental): Participants will receive 8 weeks of CBT4CBT and incentives for timely shipping. In addition, those in the CM Condition will receive at least $20 for each PEth-negative sample. Participants will receive an additional $5 for each week of consecutive negative PEth tests, with a $90 cap. In Initiation Phase, participants will attend virtual visits, provide PEth samples, and be rewarded for a decrease in PEth weekly. Maintenance Phase will begin when a participant's PEth sample is < 20 ng/mL. In Maintenance Phase, participants will attend visits and submit PEth samples every two weeks for four weeks (i.e., weeks 6 & 8). They will then attend visits and submit PEth samples every four weeks (weeks 12, 16, 20, 24), and on week 26. If participants submit a positive PEth sample, they will return to Initiation Phase and receive $20 for their next negative sample. Participants will attend visits and submit samples weekly until their PEth level is < 20 ng/mL and they restart Maintenance Phase.
  Interventions: Behavioral: Contingency Management; Behavioral: Computer Based Training for Cognitive Behavioral Therapy for AUD (CBT4CBT)

INTERVENTIONS:
Behavioral: Contingency Management — Contingency Management (CM) is an intervention that uses positive reinforcement (e.g. gift cards) to reinforce a desired behavior (e.g. negative alcohol biomarker tests) on a frequent (e.g. weekly), escalating (e.g. $5/week) schedule (e.g. 26 weeks) in order to increase the occurrence of that behavior (e.g. long term alcohol abstinence or reduction in drinking).
  Other Names: Motivational Incentives
  Arms: CM Condition (Contingency Management + CBT4CBT)
Behavioral: Computer Based Training for Cognitive Behavioral Therapy for AUD (CBT4CBT) — CBT4CBT is an evidence-based online intervention that teaches CBT principles and skills to help people with alcohol use disorder reduce their drinking. CBT4CBT teaches CBT principles through video, graphics, audio instruction, and interactive exercises. Modules include video-based examples to emphasize learning of behavioral, cognitive, and affective strategies, with an emphasis on learning from examples of individuals using skills in a range of situations. Skills taught include functional analysis, coping with craving and emotions, problem solving, decision making, challenging thoughts, and assertive alcohol refusal. Interactive exercises and homework are used to encourage skills learning and practice.

SUMMARY:
The overall objective of this program of research is to utilize phosphatidylethanol (PEth), a blood-based biomarker that can detect alcohol use for up to 28 days to deliver a feasible telehealth-based 26-week CM intervention. This study will test a telehealth PEth-based CM model in a sample of adults with AUD (n=200), recruited via online platforms by randomizing individuals to six months of 1) an online cognitive behavioral therapy for AUD (CBT4CBT) and telehealth PEth-based CM (CM condition) or 2) CBT4CBT and reinforcers for submitting blood samples (no abstinence required) (control condition). Investigators will assess group differences in PEth-defined abstinence and regular excessive drinking (PEth >= 200 ng/mL), and alcohol-related harms (e.g., smoking, drug use). This study will address important gaps in CM research by assessing outcomes during a 12-month follow-up, which is much longer than most previous CM studies; using a conceptual model to identify predictors of post-treatment abstinence. Investigators will conduct an economic analysis to place the cost of this model in the context of downstream CM-associated cost-offsets and improvements in personal and public health.

DETAILED DESCRIPTION:
The overall objective of this study is to utilize phosphatidylethanol (PEth), a blood-based biomarker that can detect alcohol use for up to 28 days to deliver a feasible telehealth-based 26-week CM intervention. In a pilot trial, we developed a telehealth-based PEth CM intervention where participants used a medical device, the TASSO-M20 to self-collect blood for PEth testing under the observation of research staff over Zoom. This intervention used a two-phase approach where the frequency of PEth testing and reinforcement was decreased from once a week, to as infrequently as every four weeks once participants achieved a PEth level consistent with two to four weeks of abstinence (< 20 ng/mL). Seventy-one percent of CM participants achieved >4 weeks of abstinence versus 21% of the treatment as usual (TAU) group, and 43% of CM participants achieved >24 weeks of abstinence compared to 0% of the TAU group (p < 0.05). Based on these promising results, this study will test a telehealth PEth-based CM model in a sample of adults with AUD (n=200), recruited via online platforms by randomizing individuals to six months of 1) an online cognitive behavioral therapy for AUD (CBT4CBT) and telehealth PEth-based CM (CM condition) or 2) CBT4CBT and reinforcers for submitting blood samples (no abstinence required) (control condition). Investigators will assess group differences in PEth-defined abstinence and regular excessive drinking (PEth >= 200 ng/mL), and alcohol-related harms (e.g., smoking, drug use). This study will address important gaps in CM research by assessing outcomes during a 12-month follow-up, which is much longer than most previous CM studies; using a conceptual model to identify predictors of post-treatment abstinence. The primary barrier to the dissemination of this model is the cost of PEth testing and CM reinforcers. Investigators will conduct an economic analysis to place these costs in the context of downstream CM-associated cost- offsets and improvements in personal and public health. If this model increases alcohol abstinence and is cost-effective it could reach millions of Americans with AUD that cannot or do not seek in-person care.

ELIGIBILITY:
Inclusion Criteria:

1. Had 2 heavy drinking episodes (assigned male at birth > 4 standard drinks (SDs), assigned female at birth > 3 SDs) or ≥14 SDs in the prior 14 days verified by PEth 16:0/18:1 biomarker > 20 ng/mL (indicates at least 2 heavy drinking episodes in past two weeks);
2. Have a DSM-5 diagnosis of a current AUD as assessed by the Structured Clinical Interview for DSM-5;
3. 18+ (individuals over 65 will be assessed for cognitive impairments)
4. Are not receiving treatment for AUD
5. Are able to complete virtual study visits via Zoom

Exclusion Criteria:

1. have a current diagnosis of severe substance use disorder (other than AUD, tobacco, and cannabis);
2. PEth biomarker ≤ 20 ng/mL (indicates no heavy drinking in past month)
3. inability to provide informed consent based on the UBACC or MacCAT-CR;
4. alcohol withdrawal-related seizure or hospitalization in prior 12 months;
5. psychiatrically or medically unsafe to participate, as assessed by the PI; and/or
6. currently enrolled in alcohol treatment or another alcohol treatment study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2028-04-04 (Estimated)

PRIMARY OUTCOMES:
Aim 1) Alcohol Abstinence & Aim 3) Predictors: PEth-Defined Alcohol Abstinence During CM (Aim 1) and Follow-Up (Aim 3) | Every study visit, up to 18 months
  Investigators will use PEth 16:0/18:1, detectable from 8 to 5,000+ ng/mL via HPLC/MS/MS to assess the primary outcome. Abstinence from alcohol, the primary outcome, will be defined as a week-over-week PEth 16:0/18:1 reduction in Initiation Phase and PEth 16:0/18:1 < 20 ng/mL in Maintenance Phase. The primary Aim 3 outcome will be PEth-defined abstinence (PEth 16:0/18:1 < 20 ng/mL) during the 12-month follow-up.
Aim 2) Alcohol-Related Harms: Addiction Severity Index (ASI) Lite | Once a month during the intervention, Follow Up, up to 18 months
  The ASI Lite will be used to assess the impact of alcohol use on psychiatric, legal, medical, and family functioning, as well as self-reported drug use.
Aim 2) Alcohol-Related Harms: Patient Health Questionnaire-9 (PHQ-9) | Once a month during the intervention, Follow Up, up to 18 months
  Depression symptoms will be assessed with the PHQ-9. Scores range from 0-27. A score of 1-4 is consistent with minimal depression, a score of 5-9 is consistent with mild depression, a score of 10-14 is consistent with moderate depression, a score of 15 to 19 is consistent with moderately severe depression, and a score of 20-27 is consistent with severe depression. Lower depression scores are treated as a better outcome.
Aim 2) Alcohol-Related Harms: Generalized Anxiety Disorder-7 (GAD-7) | Once a month during the intervention, Follow Up, up to 18 months
  Anxiety symptoms will be assessed using the GAD-7. A score of 0-4 is consistent with minimal anxiety, 5-9 with mild anxiety, 10-14 with moderate anxiety, and 15-21 with severe anxiety. A lower anxiety score is treated as a better outcome.
Aim 2) Alcohol-Related Harms: Short Form Health Survey-12 (SF-12) | Once a month during the intervention, Follow Up, up to 18 months
  Physical health will be assessed using the SF-12. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health. Higher scores will be considered a more positive outcome.
Aim 2) Alcohol-Related Harms & Aim 4) Cost Analysis: Non-study Medical and Other Services (NMOS) form | Once a month during the intervention, Follow Up, up to 18 months
  Service utilization, employment, and education will be assessed by self-report using an NMOS form. Healthcare utilization will be assessed by self-reported, time-anchoring methods. Healthcare services will include non-study: inpatient, outpatient, emergency department; SUD medications; residential and outpatient SUD treatment days; hospital detoxification days; and mental health treatment visits. This information will be gathered for the 30 days prior to baseline, then "since the last assessment." Use of non-medical and other resources required for the economic evaluation from state-policymaker and societal perspectives (e.g., criminal-legal, safety-net utilization, labor productivity, travel time to medical care) will also be collected.
Aim 2) Alcohol Related Harms: Fagerstrom | Once a month during the intervention, Follow Up, up to 18 months
  Nicotine use will be assessed using the Fagerstrom Test for Nicotine Dependence.
Aim 2) Alcohol Related Harms: Urine Drug Tests | Every study visit, up to 18 months
  Point of care urine drug test immunoassay cups will be used to assess cocaine, amphetamine, methamphetamine, cannabis, and opioid use . Participants will collect urine in the privacy of their bathroom, and display the results of their urine drug test on camera to study staff. Results are binary positive/negative for each drug class.
Aim 2) Alcohol Related Harms: Perceived Stress Scale (PSS-10) | Every study visit, up to 18 months
  Stress will be assessed with the 10-item PSS-10 to determine perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. Lower scores will be considered better outcomes.
Aim 3) Predictors: Demographics | Baseline
  Demographics, such as age, sex assigned at birth, gender, race, ethnicity, education level, housing status, and income will be assessed of predictors of alcohol use outcomes.
Aim 3) Predictors: Addictions Neuroclinical Assessment (ANA) Questionnaire | Every study visit, up to 18 months
  The ANA domains of executive functioning, negative affect, and incentive salience will be assessed via a 15-item questionnaire. Subdomains will be assessed as predictors of alcohol use outcomes.
Aim 3) Predictors: TestMyBrain | Baseline
  Performance-base measures of executive functioning, including divided attention, working memory, mental flexibility, response inhibition, impulsivity, and delay discounting will be self-administered remotely using the TestMyBrain.org platform
Aim 3) Predictors: Positive Negative Affect Schedule (PANAS) | Every study visit, up to 18 months
  Anhedonia will be measured with the 20-item PANAS. Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect. Scores will be assessed as predictors of alcohol use outcomes.
Aim 3) Predictors: Situational Confidence Questionnaire-8 (SCQ-8) | Every study visit, up to 18 months
  Alcohol Craving will be measured with the 8-item SCQ-8. Each item, representing a "situation", is scored from 0 to 100. High scores (80 and above) indicate high confidence in being able to cope with craving. Low scores (0 to 20) indicate lower confidence in coping with craving and avoiding alcohol use. A global self-efficacy score can be calculated by taking the average of all of the situations. Scores will be assessed as predictors of alcohol use outcomes.
Aim 3) Predictors: Alcohol Craving VAS | Every study visit, up to 18 months
  Alcohol Craving self-report over the past week and during the visit will be measured with a 1-100 Visual Analog Scale. A score of 0 is consistent with no alcohol craving, a score of 100 is consistent with the most alcohol craving. Scores will be assessed as predictors of alcohol use outcomes.
Aim 4) Cost Analysis: Drug Abuse Treatment Cost Analysis Program (DATCAP) | Baseline
  Resources required to implement and sustain each intervention will be identified via microcosting analysis and the DATCAP, a standardized, customizable tool that captures intervention costs in a manner conducive to estimating costs across settings.
Aim 4) Cost Analysis: PROPr | Once a month during the intervention, Follow Up, up to 18 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference (PROPr) measures a participant's health-related quality-of-life (HRQoL) across PROMIS domains of cognition, depression, anxiety, fatigue, pain interference, pain intensity, physical function, sleep disturbance, and ability to participate in social roles and activities. PROPr can generate a health utility index value, based on the participant's domain scores, that represents the US population's reference for the respondent's current health state. PROPr has five levels for each domain, ranging from "no" to "extreme" problems.

SECONDARY OUTCOMES:
Aim 1) Alcohol Abstinence: Regular excessive drinking | Every study visit, up to 18 months
  Defined as PEth 16:0/18:1 >=200 ng/mL.

OTHER OUTCOMES:
Aim 1) Alcohol Abstinence: uEtG-Defined Alcohol Abstinence | Every study visit, up to 18 months
  Urine samples will be tested for uEtG at each visit using uEtG dipcards with a threshold of 300 ng/mL
Aim 1) Alcohol Abstinence: Self-reported Alcohol Abstinence and Heavy Drinking | Every study visit, up to 18 months
  Assessed by the Alcohol Timeline Follow Back (TLFB)
Additional Implementation Data: Attrition | Every study visit, up to 18 months
  We will record attrition, defined as one month of no contact with the study team, and track attendance at study appointments.
Additional Implementation Data: CSQ-8 | Weeks 4 & 26
  To assess participant satisfaction, we will administer the 8-item Client Satisfaction Questionnaire (CSQ-8) at weeks four and 26, with a mean score of > 23 indicating overall satisfaction.
Adverse Events | Every study visit, up to 18 months
  Risks related to suicidality, dangerous alcohol use, and withdrawal symptoms will be recorded. Withdrawal symptoms will be assessed at every visit using the Sweating, Hallucinations, Orientation, Tremor (SHOT) scale, with adaptations for virtual observation and evaluation. Time spent in inpatient mental and physical health care, incarceration, visits to residential treatment programs, and other controlled environments will be recorded. Symptoms of suicidal risk will be assessed at monthly and follow-up visits.
Computer Based Training for Cognitive Behavioral Health (CBT4CBT) Program Use | Treatment & Follow up, up to 18 months
  Completion of CBT4CBT modules, scores on practice quizzes, and participant reported use of CBT4CBT skills will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonell, PhD, Principal Investigator — Washington State University Elson S. Floyd College of Medicine; Nathalie Hill-Kapturczak, PhD, Principal Investigator — University of Texas Health San Antonio; Sean Murphy, PhD, Principal Investigator — Weill Cornell
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information will be shared through the NIAAA Data Archive. Data will be linked to a GUID and include surveys, interviews, and biological test results
Supporting Information: Study Protocol
Time Frame: Data uploads to the archive will begin April 1 2024
Access Criteria: Account with the NIAAA Data Archive